CLINICAL TRIAL: NCT04665687
Title: Clinical Sequencing Project for Early Gastric Cancer and Precancerous Gastric Adenoma Patients for Personalized Cancer Clinic
Brief Title: Clinical Application of Genetic Sequencing of Early Gastric Cancer and Gastric Adenoma Patients
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyuk Lee, Samsung Medical Center, Samsung Medical Center
Other Study IDs: 2020-08-070-002
Record Dates: First submitted 2020-11-08; First posted 2020-12-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Early Gastric Cancer; Gastric Adenoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood will be collected as follows from patients with early gastric cancer or precancerous gastric adenoma that satisfy the inclusion and exclusion criteria. Tissue will be collected through biopsy/endoscopic removal peformed prior to participation in this study. Biopsies will not be performed simply for research purposes. If a biopsy is performed during the follow-up process after treatment, relevant samples will be stored if an appropriate amount of the sample remains after the biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Because advanced gastric cancer shows poor prognosis, it is important to detect early gastric cancer or precancerous gastric adenoma patients who have a cure rate of 95% or more. Moreover, a large part of early gastric cancer can be completely resected by endoscopic resection, thus ensuring a very high quality of life for patients. However, there are currently no markers that can be used for diagnosis of early gastric cancer or gastric adenoma. In addition, the biggest problem after endoscopic resection of early gastric cancer is metachronous recurrence of the cancer, which requires repeated endoscopic resection or additional surgical gastrectomy. However, there are no discovered markers for prediction of recurrence.

Liquid biopsy is a method of obtaining body fluids such as gastric juice or effusion through an endoscopic inlet during gastroscopy or colonoscopy and blood. Based on the advanced analysis method, liquid biopsy reveals more genetic information than tissue biopsy. Therefore, it is highly likely to become an essential factor in future personalized medicine. Therefore, this study was designed to identify whether tumor's molercular profiling based on tissue or blood could be used for prediction of prognosis and diagnosis of early gastric cancer and precancerous gastric adenoma.

DETAILED DESCRIPTION:
1. Acquisition of tumor samples : Tissue and 10ml of blood will be collected for genomic examination of those histologically diagnosed with early gastric cancer or precancerous gastric adenoma lesion, and additional tissue and blood will be collected at 2 months, 1 year after treatment, and recurrence.
2. Suitability of tmor samples

   : Tumor areas (> 60%) are dissected under microscopy from 4-μm-thick unstained sections by comparison with an H&E stained slide, and genomic DNA was extracted using a Qiagen DNA FFPE Tissue Kit (Qiagen, Hilden, Germany) according to the manufacturer's instructions. After extraction, we measured concentrations and 260/280 and 260/230 nm ratios using a spectrophotometer (ND1000, Nanodrop Technologies, ThermoFisher Scientific, MA, USA). Each sample was then quantified with an Qubit fluorometer (Life Technologies, Carlsbad, CA, USA). Samples of genomic DNA with more than 10 ng measured by the Qubit fluorometer were subjected to AmpliSeq library preparation. To identify "druggable" CNVs, we used a 21-gene nCounter CNV assay.
3. Method of tumor molecular profiling

   * Ion Torrent PGM Amplieq Cancer Panel 2.0 : We use the Ion AmpliSep Cancer Panel V2(Ion Torrent) to detect frequent somatic mutations that were selected based on literature review. It examines 285 mutations in 50 commonly mutated oncogenes and tumor supressor genes. First, 10ng of DNA from each 89 FFPE tumor samples underwent single-tube, multiplex PCR amplication using the Ion AmpliSepCancer Primer Pool and the AmpliSepKit reagents (Life Technologies).Treatment of the resulting amplicons with FuPa Preagent partially digest the primers and phosphorylate the amplicons. The phosphorylate the amplicons are ligated to Ion dapters and purfied. For barcoded library preparation, we substitite barcoded adapters from the Ion XpressTM Library Kit. The ligated DNA undergose nick translation and amplication to complete the linkage between adapters and amplicons and to generate sufficient material for dowmstream template treparation. Two rounds of Agencourt® AMPure® XP Reagent binding at 0.6 and 1.2 bead- to- sample volum ratios removed input DNA and unincorporated primers form the amplicons. The final library molecules are 125-300bp in size. We then transfer the libries to the Ion OneTouchTM system for automated template preparation. Sequencing is performed on the Ion PGMTM sequencer according to the manufacturer's instructions. We use IonTorrent Software for automated data analysis.
   * nCounter copy Number Variation CodeSets : We custom designed a 21-gene CNV assay as outlined in a previous study. The 21 genes included AURAKA, CCND1, CCNE1, CDK4, CDK6, CDNK1A, CDNK2A, EGFR, ERBB2, ERBB3, FGFR1, FGFR2, IGFR1R, KLF5, KRAS, MDM2, MET, MITF, MYC, PIK3CA, and TNIK. For detection of CNVs, nCounter Copy Number Variation CodeSets were used with 200 ng purified genomic DNA. DNA was fragmented via AluI digestion and denatured at 95°C. Fragmented DNA was hybridized with the codeset of 21 genes in the nCounter Cancer CN Assay Kit (Nanostring Technologies) for 18 h at 65°C and processed according to the manufacturer's instructions. The nCounter Digital Analyzer counted and tabulated the signals of reporter probes. Quantified data were analyzed using NanoString's nSolver Analysis Software.
   * Immunohistochemistry

     : RET, ATM, PD-L1, FGFR2, MLH, EGFR, ALK, ROS, TRKA. MET, HER2, PTEN loss (EGFR,CCNEI in selected cases)
   * Cancer Scan

     : targeted deep sequencing at Samsung Genome Institute

     : Illumina HiSeq2000/2500-based, MiSeq NGS targeted sequencing
   * ASFA™ Spotter
4. Statistics : Analysis of genetic research is primarily technical. Data are presented using summary statistics tables and graphs. The total disease-free survival period is calculated by the Kaplan-Meier method through medical records of subjects who have undergone endoscopic resection.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are over the age of 19
2. Those who were histologically confirmed with early gastric cancer or precancerous gastric adenoma
3. Patients with early gastric cancer or precancerous gastric adenoma falling under the above criteria who have excess tissue stored from previous non-research purpose biopsy/endodoscopic removal for treatment and diagnosis
4. Those whose life expectancy is more than 3 months
5. Those who have voluntarily consented to participate in this clinical trial

Exclusion Criteria:

1. Those who will not yield enough samples
2. Those who are considered inappropriate for this study in the discretion of the researchers

Ages: 19 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 1730 patients with early gastric cancer and precancerous gastric adenoma will be enrolled. Based on previous studies, approximately 20% of the subjects are expected to have mutations. In this study, metachronous tumor recurrence rate between the mutation group and non-mutation group will be compared. In general, metachronous tumor recurrent rate after endoscopic resection for early gastric cancer or gastric ademona is reported to be 6%-10%. In this study, the metachronous tumor recurrence rate is expected to be 10% and 5% in the mutation and non-mutation group, respectively. When a two-sided chi-square test with a power of 5% and 90% type 1 error is performed, 346 and 1384 subjected are expected to be included in the mutation group and non-mutation group, respectively.
Sampling Method: Probability Sample
Enrollment: 1730 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify biomarkers for differential diagnosis between early gastric cancer and precancerous adenoma. | From the date of initial treatment until the date of first recurrence or up to 2 years, whichever came first.
  Tumor's moleular profiling is assessed by following method:
  1. Ion Torrent PGM Amplieq Canccer Panel 2.0
  2. Nanostring copy number variation (CNV) panel
  3. Immunohistochemistry: RET, ATM, PD-L1, FGFR2, MLH, EGFR, ALK, ROS, TRKA. MET, HER2, PTEN loss (EGFR,CCNEI in selected cases)
  4. Illumina HiSeq2000/2500-based, MiSeq NGS targeted sequencing
  5. ASFA™ Spotter
Indentify prognostic biomarkers for predicting recurrence of early gastric cancer and precancerous adenoma lesion. | From the date of initial treatment until the date of first recurrence or up to 2 years, whichever came first.
  Comparison of tumor's molecular profile between the cases of recurrence and non-recurrence.
  Tumor's moleular profiling is assessed by following method:
  1. Ion Torrent PGM Amplieq Canccer Panel 2.0
  2. Nanostring copy number variation (CNV) panel
  3. Immunohistochemistry: RET, ATM, PD-L1, FGFR2, MLH, EGFR, ALK, ROS, TRKA. MET, HER2, PTEN loss (EGFR,CCNEI in selected cases)
  4. Illumina HiSeq2000/2500-based, MiSeq NGS targeted sequencing
  5. ASFA™ Spotter

SECONDARY OUTCOMES:
Change in the tumor's molecular profile on serial biopsies at the time of initial treatment, 2 months after treatment, 1 year after treatment, or recurrence. | From the date of initial treatment until the date of first recurrence or up to 2 years, whichever came first.
  The method of tumor's moleular profiling is same as the above.

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided